CLINICAL TRIAL: NCT00711607
Title: A Combined Multiple Dose and Single Dose Trial to Assess the Pharmacokinetic Profile of NOMAC, E2 and E1 After Oral Administration of NOMAC-E2 in Healthy Female Volunteers
Brief Title: A Trial to Assess the Pharmacokinetic Profile (e.g., Uptake, Distribution and Excretion of a Substance in the Body) of Nomegestrol Acetate (NOMAC), Estradiol (E2) and Estrone (E1) After Multiple and Single Dose Administration of the Combined Oral Contraception NOMAC-E2 (COMPLETED)(P05822)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: CRS Mannheim GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P05822; 292006
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: pharmacokinetics (PK); combined oral contraceptive; nomegestrol acetate; estradiol; NOMAC; E2; NOMAC-E2; pharmacokinetics
MeSH Terms: interventions — nomegestrol acetate; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group 1: NOMAC-E2 (days 1-24 and day 35)
  Interventions: Drug: nomegestrol acetate and estradiol
- 2 (Placebo Comparator): Group 2: NOMAC-E2 (days 1-24) followed by Placebo (day 35)
  Interventions: Drug: nomegestrol acetate and estradiol

INTERVENTIONS:
Drug: nomegestrol acetate and estradiol — Group 1: one tablet of 2.5 mg NOMAC-E2 and 1.5 mg E2 per day on days 1-24 and day 35; Group 2: one tablet of 2.5 mg NOMAC-E2 and 1.5 mg E2 per day on days 1-24 followed by one Placebo tablet on day 35
  Other Names: NOMAC-E2; Org 10486-0 + Org 2317

SUMMARY:
The primary purpose of this trial is to assess the pharmacokinetic profile of NOMAC, E2 and E1 after multiple and single dose administration of the combined oral contraceptive NOMAC-E2

DETAILED DESCRIPTION:
This trial was designed to assess the pharmacokinetic profile of NOMAC, E2 and E1 after multiple dose (MD) and single dose (SD) administration of NOMAC-E2 in healthy female volunteers.

In total 25 subjects were to enter the trial. These subjects were synchronized for menstrual cycle by taking 1 tablet NOMAC-E2 (2.5 mg / 1.5 mg) daily for a minimum of 2 weeks. This was followed by a 7-day pill-free interval. After this, all subjects were to be exposed to the open-label MD treatment with 1 tablet NOMAC-E2 (2.5 mg / 1.5 mg) once daily, during 24 days. This was followed by a second pill-free interval of 10 days, to allow for sufficient washout of NOMAC-E2. On treatment day 35, 20 subjects were to receive 1 tablet NOMAC-E2 (2.5 mg / 1.5 mg) and 5 subjects were to receive a placebo tablet in a double blinded setup. After treatment day 35 and before follow-up, all subjects would again have a pill-free interval of 7 days. After follow-up, all subjects could return to their own contraceptive schedule. Follow-up took place on treatment day 42.

Bleeding pattern and tablet intake were assessed by means of a subject diary to be completed on a daily basis. Blood sampling for pharmacokinetic and pharmacodynamic purposes were collected at several time points before, during and after the MD and SD period. In order to explore any possible influence of NOMAC-E2 on the QT/QTc interval, a small placebo group was designed within the SD period, to allow for comparison with the active-treated group. In addition several safety assessments (vital signs, ECGs, trans vaginal ultrasound evaluation, physical, gynecological and breast examinations, cervical smear, routine laboratory parameters and adverse events) were performed.

ELIGIBILITY:
Inclusion Criteria:

* Fertile female subjects in good physical and mental health and 18 - 50 years of age at screening
* Body mass index (BMI) of 17 ≤ BMI ≤ 29 kg/m2
* Able and willing to use non-hormonal contraceptives during the trial from screening up to follow up
* With the last menstrual cycle of 28 +/- 7 days
* Able and willing to sign the informed consent form
* Able to refrain from smoking, grapefruit containing products, and all use of (methyl)xanthines (e.g. coffee, tea, cola, chocolate) during hospitalization and during pharmacokinetic sampling on days 24-30 and days 35-41

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to NOMAC-E2 or chemically related compounds or excipients which could be employed within the study or to any other unknown drug used in the past
* Use of any drug or substance within one week prior to the first treatment day, except paracetamol
* Clinically relevant history or presence of any medical disorder
* Clinically relevant abnormal laboratory, ECG, vital signs or physical findings at screening (and just prior to dosing)
* Known or suspected pregnancy
* History of/or current abuse of drugs or alcohol or solvents, or positive drug or alcohol screen at screening and admission, as judged by the investigator
* Positive test result on hepatitis B surface antigen, hepatitis C antibody, or HIV 1/2 serology
* Participation in an investigational drug study within 90 days prior to treatment day 1
* Donation of blood within 90 days prior to treatment day 1
* Contra-indications of contraceptive steroids (general)
* Abnormal cervical smear at screening, or documentation of abnormal smear performed within 12 months before screening
* Clinically relevant transvaginal ultrasound pathology or inability to undergo transvaginal ultrasound evaluation
* Use of an injectable hormonal method of contraception; within 6 months of an injectable with a 3-month duration, within 4 months of an injectable with a 2-month duration, within 2 months of an injectable with a 1-month duration
* Before spontaneous menstruation has occurred following a delivery or abortion
* Breastfeeding or within 2 months after stopping breast feeding prior to start of trial medication
* Present use or use during two months prior to the start of the trial medication of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex steroids (other than pre- and post treatment contraceptive method) and herbal remedies containing hypericum perforatum (St. John's Wort)
* Present use or use within one month prior to screening of any agent that was known to prolong the QT/QTc interval
* History of /or current risk factors for TdP (e.g. heart failure, hypokaliemia, hypomagnesaemia, hypocalcaemia, family history of long QT syndrome, loss of consciousness)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2007-09-01 (Actual); Study Completion 2007-09-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of NOMAC and serum concentrations of E2 and E1 measured at several time points before, during and after multiple dose and after single dose administration to determine pharmacokinetics | days 1 to 24, and days 34 - 42

SECONDARY OUTCOMES:
Time-matched mean effects of QTcB, QTcF and QTcI values (respectively Bazett, Fredericia and Individual correction methods) compared to placebo, and time-matched changes from baseline | Screening (week -5), days 34, 35 and 42;
Drug safety as determined by gynecological and breast examination, trans vaginal ultrasound evaluation, pregnancy test, vital signs, ECG recordings, adverse events monitoring, routine laboratory parameters | From week -5 (screening) upto and including day 42 (followup)
Pharmacodynamics as determined by measuring serum concentrations of progesterone, luteinizing hormone (LH), follicle stimulating hormone (FSH) and sex hormone binding globulin (SHBG) | days 1 to 24, and days 34 - 42

REFERENCES:
- [Result] Gerrits MG, Schnabel PG, Post TM, Peeters PA. Pharmacokinetic profile of nomegestrol acetate and 17beta-estradiol after multiple and single dosing in healthy women. Contraception. 2013 Feb;87(2):193-200. doi: 10.1016/j.contraception.2012.07.001. Epub 2012 Aug 13. PMID 22898360